CLINICAL TRIAL: NCT07181876
Title: Robotic Minimally Invasive Inguinal Hernia Repair Post-Market Clinical Study With the DEXTER Robotic System
Acronym: RAS-ACCESS
Status: Recruiting | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Veranex, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-03
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Inguinal Hernia Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: inguinal hernia repair — Robotic-assisted inguinal hernia repair with the DEXTER robotic surgery system

SUMMARY:
The purpose of this post-market, observational study is to collect data under anticipated conditions of use that demonstrates that DEXTER performs as intended in the intended patient population, including a variety of representative disease etiologies and demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 22 years of age at time of enrollment/consent
* Subject is indicated for and planned to undergo robot-assisted and laparoscopic surgery for unilateral or bilateral inguinal hernia repair
* Subject is able and willing to comply with the protocol requirements, has been informed of the nature of the study, and has signed the IRB-approved informed consent form

Exclusion Criteria:

* Subject with any relative and absolute contraindications for the use of conventional endoscopes and endoscopic surgical instruments and/or general non-procedure specific contraindications to endoscopic surgery including bleeding diathesis and pregnancy
* Subject is participating in another clinical investigation at the time of enrollment or planned participation at any time during this clinical study
* Subject has a known or suspected medical condition that, in the opinion of the Investigator, may put the subject at risk for participation in this clinical study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing unilateral or bilateral inguinal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary safety outcome | up to 30 days after surgery
  Occurrence of Clavien-Dindo grades III-V adverse events
Primary efficacy outcome | Intraoperative
  Successful completion of the DEXTER-assisted procedure, i.e. free of any conversion to an open or fully laparoscopic surgical approach

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northtowns Ambulatory Surgical Center (NASC), Buffalo, New York
  - Memorial Hermann-Texas Medical Center - UT Health Houston, Houston, Texas